CLINICAL TRIAL: NCT06619197
Title: Exploratory Study on Global Reflexology Proposed in the Management of Pain in Children With Sickle Cell Disease in Vaso-occlusive Crisis
Brief Title: Exploratory Study on Global Reflexology in Sickle Cell Disease
Acronym: REFLEXODREPANO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL22_0315; 2023-A01667-38 (Other: ID-RCB)
Record Dates: First submitted 2024-09-13; First posted 2024-10-01 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Reflexology; Pain; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Intervention Model Description: Prospective exploratory study of single-center feasibility. Research involving human subjects 2. This feasibility study will estimate the improvement in pain provided by reflexology, acceptability and feasibility, rate of inclusion.
  The research will take place in 2 centers, the short-stay hospitalization unit (UHCD) and the continuous monitoring unit (USC) of the Women's Mother and Child Hospital of the Hospices Civils de Lyon.
  This study involves subjects under 18 years of age, suffering from sickle cell disease, hospitalized in the unit UHCD or the unit USC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- global reflexology (Other): This study involves subjects under 18 years of age, suffering from sickle cell disease, hospitalized in the short-stay hospitalization unit (UHCD) or continuous monitoring unit (USC) of the Women's Mother and Child Hospital of the Hospices Civils de Lyon.
  Interventions: Other: Global reflexology

INTERVENTIONS:
Other: Global reflexology — The EMC method is a global reflexology technique inspired by the work of the American naturopath Stanley Burrough (Vitaflex, 1976). It is a method of reflexology on the whole body, of acupressure massages (rhythmic and targeted movements) on so-called "reflex" zones which is practiced on different areas of the body (feet, hands, arms, legs, collarbone, ear) and allows the stimulation of all systems.

SUMMARY:
Sickle cell disease (or sickle cell anemia) is the most common genetic disease in France with 586 children screened in 2019. This chronic disease is characterized by the presence of abnormal Hemoglobin (Hb) S and a deformation of the red blood cells which take the elongated shape of a sickle and become more rigid and more fragile. Sickle cell disease manifests itself among other things by very painful vaso-occlusive crises (VOC) and for some chronic pain.

Their management is an emergency and often requires hospitalization. Despite analgesic treatment, some patients have persistent pain.

In 2013, a childcare assistant trained in Canadian global reflexology EMC offered reflexology sessions to 12 sickle cell patients. She observed a relief in all patients with a decrease in the pain score in 8 of them. These sessions seem to show us a double interest: the reduction of the child's pain and the emergence of a technique that can be used by paramedics in the context of their own role.

The investgators hypothesize that global reflexology is an effective and acceptable complementary technique for pain management in addition to the usual analgesic management in sickle cell children under 18 years of age in CVO. In order to verify our hypothesis, the investigators propose to explore the practice of Canadian global reflexology as an innovative therapeutic option complementary to drug treatments in the hospital management of sickle cell children.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 years of age
* Patient suffering from sickle cell disease
* Patient hospitalized in the UHCD or USC unit of the Women's Mother and Child Hospital of the Hospices Civils de Lyon for the management of a CVO
* Informed consent signed by at least one holder of parental authority
* Collection of the patient's assent as soon as his age allows it.

Exclusion Criteria:

* Patient with PCA (Patient Controlled Analgesia)
* Patient with NCA (Nurse Controlled Analgesia)
* Patient not affiliated to a social security scheme or beneficiaries of a similar scheme.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain score T20 with the Face Legs Activity Cry Consolability scale | 20 minutes after the start of the session
  Evolution of pain scores (Face Legs Activity Cry Consolability - FLACC according to the child's age) T0 and T20 minutes after the start of the session.
  The minimum value is 0 (no pain) and the maximum is 10 (maximum pain). All professionals are trained in the use of the FLACC pain scale
Pain score T20 with the Visual Analog Scale | 20 minutes after the start of the session
  Evolution of pain scores (VAS - Visual Analog Scale according to the child's age) T0 and T20 minutes after the start of the session. The minimum value is 0 (no pain) and the maximum is 10 (maximum pain). All professionals are trained in the use of the VAS pain scale

SECONDARY OUTCOMES:
Pain score T80 with the Visual Analog Scale | 80 MINUTES after the start of the session
  Changes in pain scores (VAS - Visual Analog Scale according to the child's age) at each session between T0 and T80 minutes after the start of the session. The minimum value is 0 (no pain) and the maximum is 10 (maximum pain). All professionals are trained in the use of the VAS pain scale
Pain score T80 with the Face Legs Activity Cry Consolability scale | 80 minutes after the start of the session
  Changes in pain scores (Face Legs Activity Cry Consolability according to the child's age) at each session between T0 and T80 minutes after the start of the sessionmn. The minimum value is 0 (no pain) and the maximum is 10 (maximum pain). All professionals are trained in the use of the FLACC pain scale
Length of hospitalization | 1 Month
  Length of stay of patients included in the study, defined by the time between their entry into the UHCD or USC and their return home.
Number of reflexology sessions | 1 Month
  Total number of global reflexology sessions performed for each child included in the study.
Recorded side effects, complications | 1 Month
  Recorded side effects, complications
Acceptability of the technique : refusal to participate. | 25 Months
  Acceptability of the technique: number of refusals to participate in the protocol during the study.
Acceptability of the technique: reason for refusal to participate. | 25 months
  Acceptability of the technique: reasons of refusals to participate in the protocol during the study.
Acceptability of the technique: interruption of participation. | 25 months
  Acceptability of the technique: number of requests for interruption during the study.
Acceptability of the technique: reason for interruption of participation | 25 months
  Acceptability of the technique: reasons for discontinuations for requests of interruption during the study.
Feasibility of the technique | 25 months
  Feasibility of the technique: integration into the management of CVO: number of sessions not performed or interrupted and reasons, duration of sessions.
Inclusion rate | 25 months
  Monthly inclusion rate in the study, characteristics of the eligible population, included and not included.

CONTACTS AND LOCATIONS:
Overall Officials: COLLOT SOPHIE, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France